CLINICAL TRIAL: NCT01770236
Title: Optimal Method of Pain Control After Minimally Invasive Coronary Artery Bypass Grafting
Brief Title: Pain Control After Minimally Invasive Coronary Artery Bypass Grafting
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study medication no longer available at institution
Sponsor: Gundersen Lutheran Medical Foundation (Other)
Responsible Party: Principal Investigator, Kara Kallies, Academic researcher, on behalf of PI, Prem Rabindra, MD, Gundersen Lutheran Medical Foundation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2-12-12-001
Record Dates: First submitted 2013-01-14; First posted 2013-01-17 (Estimated); Last update posted 2016-12-21 (Estimated); Status verified 2016-12

CONDITIONS: Postoperative Pain; Medication Side Effects; Narcotic Requirement
MeSH Terms: conditions — Pain, Postoperative; Drug-Related Side Effects and Adverse Reactions | interventions — Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IV acetaminophen (Experimental): Patients in this group will receive intraoperative intercostal block + IV acetaminophen (1000 mg every 6 hours for adults and weight-based for any patient under 50 kg)
  Interventions: Drug: IV acetaminophen
- On-Q Pain Pump catheter (No Intervention): Patients in this group will receive the current standard care which includes an intraoperative intercostal block + On-Q Pain Pump catheter (continuous dosing).

INTERVENTIONS:
Drug: IV acetaminophen — Patients randomized to the IV acetaminophen group will receive IV acetaminophen (1000 mg every 6 hours for adults and weight-based for any patient under 50 kg)instead of an On-Q pain pump catheter.
  Other Names: Tylenol; Ofirmev
  Arms: IV acetaminophen

SUMMARY:
The purpose of this study is to compare postoperative pain control after minimally invasive coronary artery bypass grafting for patients who receive an intercostal block (an anesthetic medicine injected in an area under the ribs) in the operating room and IV acetaminophen (Tylenol) to those who receive an intercostal block and On-Q pain pump catheter (a balloon pump attached to 2 small tubes near your procedure site that automatically delivers pain medicine).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Coronary artery disease requiring surgical intervention
* No prior sternotomy
* Creatinine within normal limits (0.60 - 1.10 mg/dL)

Exclusion Criteria:

* Less than 18 years of age
* Inability to provide consent or complete a written survey
* Previous history of sternotomy
* Contraindications to MICS-CABG or to any of the components of the 2 analgesic regimens

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2013-01; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Pain score | Participants will be followed for the duration of hospital stay, an expected average of 4 days
  Pain scores will be assessed using a Numerical Rating Scale (NRS) (an 11-point scale, 0 through 10, with 0 representing 'No pain' and 10 representing 'Worst imaginable pain'). Pain scores will be entered by nursing staff every 2 hours in ICU, and every 6 hours on the floor for the duration of the hospital stay, an expected average of 4 days.

SECONDARY OUTCOMES:
Medication side effects | Participants will be followed for the duration of hospital stay, an expected average of 4 days
  Any side effects and need for additional narcotic medication will be collected throughout the duration of the hospital stay, an expected average of 4 days.

CONTACTS AND LOCATIONS:
Overall Officials: Prem Rabindra, MD, Principal Investigator — Gundersen Health System; Kym Culp, MD, Principal Investigator — Gundersen Health System; Korey Zellner, PA-C, Principal Investigator — Gundersen Health System
Locations (1):
- Gundersen Lutheran Health System, La Crosse, Wisconsin, United States

REFERENCES:
- [Background] Walther T, Falk V, Metz S, Diegeler A, Battellini R, Autschbach R, Mohr FW. Pain and quality of life after minimally invasive versus conventional cardiac surgery. Ann Thorac Surg. 1999 Jun;67(6):1643-7. doi: 10.1016/s0003-4975(99)00284-2. PMID 10391268
- [Background] McGinn JT Jr, Usman S, Lapierre H, Pothula VR, Mesana TG, Ruel M. Minimally invasive coronary artery bypass grafting: dual-center experience in 450 consecutive patients. Circulation. 2009 Sep 15;120(11 Suppl):S78-84. doi: 10.1161/CIRCULATIONAHA.108.840041. PMID 19752390
- [Background] Berger MM, Berger-Gryllaki M, Wiesel PH, Revelly JP, Hurni M, Cayeux C, Tappy L, Chiolero R. Intestinal absorption in patients after cardiac surgery. Crit Care Med. 2000 Jul;28(7):2217-23. doi: 10.1097/00003246-200007000-00006. PMID 10921543